CLINICAL TRIAL: NCT07107802
Title: A Phase 1, Single Ascending Dose Study, to Assess the Safety and Pharmacokinetics of Intravenous ATX101 in Healthy Participants
Brief Title: Phase 1 Single Ascending Dose Study With ATX101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aurobac Therapeutics SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ATX101-CLN-1001; 2025-521999-56-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-25; First posted 2025-08-06 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ATX101 - low dose (Experimental)
  Interventions: Drug: ATX101
- ATX101 - middle dose (Experimental)
  Interventions: Drug: ATX101
- ATX101 - high dose (Experimental)
  Interventions: Drug: ATX101
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATX101 — Single intravenous dose
  Arms: ATX101 - high dose; ATX101 - low dose; ATX101 - middle dose
Drug: Placebo — Single intravenous dose
  Arms: Placebo

SUMMARY:
The main objective of this study is to assess the safety and tolerability of intravenously administered ATX101 in healthy adults following single ascending doses of ATX101. The pharmacokinetic profile of ATX101 and its metabolites will also be investigated.

DETAILED DESCRIPTION:
This is a single-center, double-blinded, placebo-controlled, phase I, single ascending dose study in healthy participants. A maximum of three ATX101 dose levels are pre-planned to be investigated in three separate sequential cohorts. Each of these cohorts will consist of 8 healthy participants (6 participants randomized to ATX101 and 2 to placebo). The study will consist of:

* a screening period, within 7 to 21 days before investigational product administration (Day -21 to Day -7),
* a treatment period, including admission to confinement, 3-night confinement, and discharge from confinement.
* a follow-up period, which includes two ambulatory follow-up visits (Day 4 and Day 7).

Total duration of study participation for each participant will be approximately 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Free written informed consent prior to any procedure required by the study.
2. Male or female participant ≥18 and ≤50 years-old, at the time of signing the informed consent.
3. Body mass index (BMI) between 18.5 and 29.9 kg/m2 and a minimum weight of 48 kg for women and 50 kg for men and maximum weight of 100 kg (inclusive).
4. No clinically relevant diseases captured in medical history.
5. No clinically relevant abnormalities at screening and admission.
6. Negative test results for anti-Human Immunodeficiency virus 1 and 2 antibodies (anti-HIV-1Ab and anti-HIV-2Ab), Hepatitis B surface antigen (HBsAg), and anti-Hepatitis C virus antibodies (anti-HCVAb).
7. A female participant is either be of non-childbearing potential; or using an accepted contraceptive method.

Exclusion Criteria:

1. Previous exposure to ATX101 or to ATX101 drug substance.
2. Known hypersensitivity/allergic reaction to the study drug substance or any of the excipients.
3. Known severe hypersensitivity reaction to any other drug.
4. If woman, she is breast-feeding.
5. Rest systolic blood pressure (SBP) <90 mmHg or >140 mmHg.
6. Rest diastolic blood pressure (DBP) <50 mmHg/or >95 mmHg.
7. Resting heart rate outside the range of 50 to 90 bpm, in the ECG.
8. Hematological and biochemistry parameters outside the normal range.
9. Renal function outside normal range.
10. Positive result in drugs-of-abuse or ethanol tests.
11. If woman of childbearing potential (WOCBP), positive pregnancy test.
12. Use of a depot injection or an implant of any drug within the previous 6 months.
13. Average weekly alcohol consumption of >14 units for males and >7 units for females, within the previous 6 months.
14. Average daily consumption of methylxanthines-containing beverages or food (e.g., coffee, tea, cola, sodas, chocolate) equivalent to >500 mg of methylxanthines, within the previous 6 months.
15. Participation in any interventional clinical trial within the previous 2 months.
16. Participation in more than 2 clinical trials within the previous 12 months.
17. Blood donation or significant blood loss (≥450 mL) due to any reason or had plasmapheresis within the previous 2 months.
18. Any other condition that the Investigator considers to render the participant unsuitable for the study.
19. Any recent disease or condition or treatment that, according to the Investigator, would put the participant at undue risk due to study participation or occurred at a timeframe in which may interfere with the pharmacokinetics of study drug.
20. Fever (≥38 ºC) in the previous week.
21. Use of prescription or nonprescription medicinal products, vitamins, food supplements or herbal supplements (including St John's Wort) within 2 weeks prior to admission to the study, unless in the Investigator's opinion the medication does not interfere with the pharmacokinetics of study drug or compromise participant safety.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-07-19 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Number and proportion of subjects with treatment-emergent adverse events (TEAEs). Occurrence of clinically relevant abnormalities on physical examination, safety laboratory tests, electrocardiogram parameters, and vital signs. | Up to Day 7

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) of ATX101 in plasma | Up to Day 4
Time of occurrence of the maximum observed concentration (tmax) of ATX101 in plasma | Up to Day 4
Area under the concentration-time curve (AUC) of ATX101 in plasma from the start of infusion (t=0h) up to the end of infusion (AUC0-T) | Up to Day 4
Partial area under the concentration-time curve (AUC) of ATX101 in plasma from the start of infusion (t=0h) up to 24 hours after the start of infusion (AUC0-24) | Up to 24 hours
Area under the concentration-time curve (AUC) of ATX101 in plasma from the start of infusion (t=0h) up to the time of last measurable concentration (AUC0-t) | Up to Day 4
Area under the concentration-time curve (AUC) of ATX101 in plasma from the start of infusion (t=0h) extrapolated to infinity (AUC0-∞) | Up to Day 4
Residual area or percentage of extrapolated part of area under the concentration-time curve of ATX101 in plasma from the start of infusion (t=0h) extrapolated to infinity (%AUCextrap) | Up to Day 4
Apparent terminal elimination rate constant (λz) of ATX101 in plasma | Up to Day 4
Apparent terminal elimination half-life (t½) of ATX101 in plasma | Up to Day 4
Apparent volume of distribution (VD) of ATX101 in plasma | Up to Day 4
Apparent total body clearance (CL) of ATX101 in plasma | Up to Day 4

OTHER OUTCOMES:
Maximum observed concentration (Cmax) of ATX101 metabolites in plasma | Up to Day 4
Time of occurrence of the maximum observed concentration (tmax) of ATX101 metabolites in plasma | Up to Day 4
Area under the concentration-time curve (AUC) of ATX101 metabolites in plasma from the start of infusion (t=0h) up to the end of infusion (AUC0-T) | Up to Day 4
Partial area under the concentration-time curve (AUC) of ATX101 metabolites in plasma from the start of infusion (t=0h) up to 24 hours after the start of infusion (AUC0-24) | Up to 24 hours
Area under the concentration-time curve (AUC) of ATX101 metabolites in plasma from the start of infusion (t=0h) up to the time of last measurable concentration (AUC0-t) | Up to Day 4
Area under the concentration-time curve (AUC) of ATX101 metabolites in plasma from the start of infusion (t=0h) extrapolated to infinity (AUC0-∞) | Up to Day 4
Residual area or percentage of extrapolated part of area under the concentration-time curve of ATX101 metabolites in plasma from the start of infusion (t=0h) extrapolated to infinity (%AUCextrap) | Up to Day 4
Apparent terminal elimination rate constant (λz) of ATX101 metabolites in plasma | Up to Day 4
Apparent terminal elimination half-life (t½) of ATX101 metabolites in plasma | Up to Day 4
Metabolic ratios (MR) estimated for ATX101 metabolites in plasma | Up to Day 4

CONTACTS AND LOCATIONS:
Locations (1):
- BlueClinical Phase I, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No
This is a healthy volunteer study being conducted to define the safety and pharmacokinetic profile of the tested drug. This study is not exploring the activity of our drug in the target indication population. As such, we do not believe there is utility for sharing deidentified IPD from this trial with other researchers.